CLINICAL TRIAL: NCT01396278
Title: A Randomised, Double-blind, Double-dummy, Active-controlled, Parallel-group Study to Assess and Compare Efficacy and Safety of an 8-week Treatment With BI 54903 at Doses of 90.9, 181.8 and 363.6 µg b.i.d. Administered Via Respimat® Inhaler and Fluticasone Propionate HFA MDI 440 µg b.i.d. in Patients With Asthma Inadequately Controlled on Medium Dose ICS Therapy
Brief Title: Study on BI 54903 (Inhaled Corticosteroid) Administered Twice Daily Via Respimat Inhaler in Patients With Asthma Inadequately Controlled on Medium Dose Inhaled Corticosteroid (ICS).
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1248.7; 2010-023169-23 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-07-15; First posted 2011-07-18 (Estimated); Results first posted 2022-06-23 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone

ARMS (5):
- BI 54903 low dose (Experimental): patient to receive Respimat inhaler containing low dose BI 54903 plus placebo matching hydrofluoroalkane (HFA) metered dose inhaler (MDI)
  Interventions: Drug: Placebo; Drug: BI 54903
- BI 54903 medium dose (Experimental): Respimat inhaler containing medium dose BI 54903 plus placebo matching HFA MDI
  Interventions: Drug: Placebo; Drug: BI 54903
- BI 54903 high dose (Experimental): Respimat inhaler containing high dose BI 54903 plus placebo matching HFA MDI
  Interventions: Drug: Placebo; Drug: BI 54903
- Fluticasone propionate 440 mcg BID (Active Comparator): Fluticasone HFA MDI containing 440 mcg ICS plus placebo matching Respimat inhaler
  Interventions: Drug: Fluticasone propionate
- Fluticasone propionate 88 mcg BID (Active Comparator): Fluticasone HFA MDI containing 88 mcg ICS plus placebo matching Respimat inhaler
  Interventions: Drug: Fluticasone propionate

INTERVENTIONS:
Drug: Placebo — Placebo matching fluticasone propionate HFA MDI
  Arms: BI 54903 high dose; BI 54903 low dose; BI 54903 medium dose
Drug: Fluticasone propionate — Fluticasone propionate HFA MDI
  Arms: Fluticasone propionate 440 mcg BID; Fluticasone propionate 88 mcg BID
Drug: BI 54903 — BI 54903 via Respimat inhaler
  Arms: BI 54903 high dose; BI 54903 low dose; BI 54903 medium dose

SUMMARY:
The aim of the study is to assess and compare efficacy and safety of BI 54903 at three different dosages (b.i.d)., fluticasone propionate hydrofluoroalkane (HFA) metered dose inhaler (MDI) at a dose of 440 mcg b.i.d and low dose fluticasone propionate 88 mcg b.i.d. over an 8-week treatment period in asthmatic patients aged 12 to 65 years inadequately controlled medium dose ICS therapy as demonstrated by a decrease in forced expiratory volume in one second (FEV1) range 10 to 25 % and an asthma control questionnaire-6 (ACQ-6) equal or greater than 1.5 at time of randomisation.

ELIGIBILITY:
Inclusion criteria:

1. Must be willing and able to give informed consent.
2. Male and female patients aged at least 12 to 65 years.
3. All patients must have a history of asthma diagnosed by a physician for at least three months at the time of enrolment into the trial according to the 2009 Global Initiative for Asthma (GINA) Guidelines. The initial diagnosis of asthma must have been made before the age of 40 years.
4. All patients must be on a maintenance treatment with high-dose ICS with long-acting beta 2-agonist (LABA), stable for at least six weeks prior to Visit 1
5. All patients must have a pre-bronchodilator FEV1 of not less than 60 to 90% of predicted normal and an ACQ-6 mean score of less than 1.5 at the pre-screening Visits 1and 2.
6. Patients must be never-smokers or ex-smokers with a smoking history of less than 10 pack-years and smoking cessation at least one year prior to screening .
7. Patients must be able to use Respimat® inhaler and MDI correctly
8. Patients must be able to perform all trial-related procedures including technically acceptable pulmonary function tests and electronic peak expiratory flow (PEF) measurements, and must be able to maintain records during the study period as required in the protocol.

   To enter treatment period following additional criteria have to be met:
9. All patients must have an improvement in FEV1 not less than 12 % above baseline and an absolute change of at least 200 mL within 15-30 min after administration of 400 mcg salbutamol/albuterol HFA MDI as demonstrated at Visit 1 or during one of the visits during run-in period.
10. During the run-in period (at the same clinic visit) all patients must be both symptomatic (ACQ-6 mean score equal to or greater than 1.5) and have shown a decrease in morning pre-bronchodilator FEV1 not less than 10% and less than or equal to 25% from pre-screening baseline FEV1 at Visit 2.

Exclusion criteria:

1. Patients with significant pulmonary disease other than asthma or other significant medical conditions (as determined by medical history, examination and clinical investigations at screening) that may, in the opinion of the investigator, result in any of the following: (i) put the patient at risk because of participation in this trial or (ii) influence the results of the trial or (iii) cause concern regarding the patient´s ability to participate in the trial.
2. Patients with a clinically relevant, abnormal screening haematology and/or blood chemistry finding, if the abnormality indicates a significant disease as defined in exclusion criterion no. 1.
3. Patients with a history of upper respiratory tract infection (URTI) or lower respiratory tract infection (LRTI) in the past four weeks prior to the pre-screening Visit 1, and during pre-screening and run-in periods.
4. Patients with any exacerbation of their underlying asthma during the eight weeks prior to the pre-screening Visit 1.
5. Patients with active allergic rhinitis requiring treatment with systemic corticosteroids.
6. Any of the following criteria are met during the pre-screening/run-in period (Visits 1 - 6):

   * in clinic pre-bronchodilator FEV1 % predicted less than 40%,
   * more than 12 puffs rescue salbutamol/albuterol HFA MDI per day for > 2 consecutive days,
   * exacerbation of asthma.
7. Patients with a history of pneumonectomy or who are planning to undergo thoracotomy for any reason.
8. Patients who are currently in a pulmonary rehabilitation program or have completed a pulmonary rehabilitation program in the six weeks prior to the first screening visit 1.
9. Patients with two or more hospitalizations for asthma within the previous 12 months.
10. Patients with a recent history of myocardial infarction during the last twelve months or known coronary heart disease that requires treatment
11. Patients with a history of hospitalisation due to heart failure in the past twelve months
12. Patients with myocarditis or any unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year
13. Patients with significant alcohol or drug abuse in the opinion of the investigator within the past two years
14. Patients with rheumatoid arthritis or other systemic diseases that require immune system modulating treatment
15. Patients suffering from or with a history of glaucoma, increased intraocular pressure, and/or cataracts
16. Pregnant or nursing women
17. Women of childbearing potential not using a highly effective method of birth control.
18. Patients who have been treated with anti-IgE-antibodies (e.g. omalizumab, Xolair®) or other immune system modulating antibodies such as tumor necrosis factor-alpha blockers (TNF-alpha blockers) within six months prior to Visit 1.
19. Patients who have been treated with the following drugs during the past four weeks prior to Visit 1 or are foreseen to need this during the study:

    * Non-selective ß-blockers (topical cardio-selective beta-blocker eye medications for non-narrow angle glaucoma are allowed),
    * Oral or other systemic corticosteroids,
    * Oral beta-agonists,
    * Changes in allergen desensitisation therapy in last 6 months,
    * Immune system modulating agents such as methotrexate or cyclosporine,
    * Inhibitors of cytochrome P450 3A4 such as antifungals (e.g. ketoconazole, itraconazole), antibiotics (e.g. erythromycin) or antiretroviral drugs.
20. Patients who have been treated with leukotriene modifiers, chromones or theophylline within two weeks prior to Visit 1.
21. Patients who have been treated with tiotropium within 3 weeks prior to Visit 1.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2011-12-01 (Actual); Study Completion 2011-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (37):
- United States (37):
  - 1248.7.01047 Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - 1248.7.01023 Boehringer Ingelheim Investigational Site, Fullerton, California
  - 1248.7.01038 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1248.7.01004 Boehringer Ingelheim Investigational Site, Mission Viejo, California
  - 1248.7.01028 Boehringer Ingelheim Investigational Site, Palmdale, California
  - 1248.7.01044 Boehringer Ingelheim Investigational Site, Stockton, California
  - 1248.7.01015 Boehringer Ingelheim Investigational Site, Centennial, Colorado
  - 1248.7.01035 Boehringer Ingelheim Investigational Site, Aventura, Florida
  - 1248.7.01022 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1248.7.01051 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 1248.7.01052 Boehringer Ingelheim Investigational Site, Savannah, Georgia
  - 1248.7.01011 Boehringer Ingelheim Investigational Site, Eagle, Idaho
  - 1248.7.01055 Boehringer Ingelheim Investigational Site, Oak Lawn, Illinois
  - 1248.7.01019 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1248.7.01039 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1248.7.01037 Boehringer Ingelheim Investigational Site, Ypsilanti, Michigan
  - 1248.7.01056 Boehringer Ingelheim Investigational Site, Rolla, Missouri
  - 1248.7.01036 Boehringer Ingelheim Investigational Site, Warrensburg, Missouri
  - 1248.7.01020 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1248.7.01049 Boehringer Ingelheim Investigational Site, Berlin, New Jersey
  - 1248.7.01026 Boehringer Ingelheim Investigational Site, Ocean City, New Jersey
  - 1248.7.01054 Boehringer Ingelheim Investigational Site, Trenton, New Jersey
  - 1248.7.01031 Boehringer Ingelheim Investigational Site, High Point, North Carolina
  - 1248.7.01045 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1248.7.01021 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1248.7.01013 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1248.7.01040 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1248.7.01012 Boehringer Ingelheim Investigational Site, Upland, Pennsylvania
  - 1248.7.01048 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1248.7.01050 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1248.7.01002 Boehringer Ingelheim Investigational Site, Live Oak, Texas
  - 1248.7.01032 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1248.7.01046 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1248.7.01001 Boehringer Ingelheim Investigational Site, Waco, Texas
  - 1248.7.01025 Boehringer Ingelheim Investigational Site, Murray, Utah
  - 1248.7.01053 Boehringer Ingelheim Investigational Site, Alexandria, Virginia
  - 1248.7.01030 Boehringer Ingelheim Investigational Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized, double-blind, double-dummy, active-controlled, parallel group study was to assess and compare efficacy and safety of an 8-week treatment with BI 54903 administered via Respimat® inhaler and fluticasone propionate hydrofluoroalkane Metered dose inhaler in patients with asthma.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 54903 90.9μg Bid: 2 puffs (total 90.9 microgram (μg)) of BI 54903 ethanolic solution for inhalation were inhaled orally via Respimat® inhaler (combined with placebo hydrofluoroalkane (HFA) Metered dose inhaler (MDI), 2 puffs twice daily (bid) in the morning and evening for a treatment period of 8 weeks.
- BI 54903 181.8μg Bid: 2 puffs (total 181.8 microgram (μg)) of BI 54903 ethanolic solution for inhalation were inhaled orally via Respimat® inhaler (combined with placebo hydrofluoroalkane (HFA) Metered dose inhaler (MDI), 2 puffs twice daily (bid)) twice daily in the morning and evening for a treatment period of 8 weeks.
- BI 54903 363.6μg Bid: 2 puffs (total 363.6 microgram (μg)) of BI 54903 ethanolic solution for inhalation were inhaled orally via Respimat® inhaler (combined with placebo hydrofluoroalkane (HFA) Metered dose inhaler (MDI), 2 puffs twice daily (bid)) twice daily in the morning and evening for a treatment period of 8 weeks.
- Fluticasone Propionate 88μg Bid: 2 puffs (total 88 microgram (μg)) of fluticasone propionate were inhaled orally from hydrofluoroalkane (HFA) Metered dose inhaler (MDI) (combined with placebo Respimat® inhaler) twice daily (bid) in the morning and evening for a treatment period of 8 weeks.
- Fluticasone Propionate 440μg Bid: 2 puffs (total 440 microgram (μg)) of fluticasone propionate were inhaled orally from hydrofluoroalkane (HFA) Metered dose inhaler (MDI) (combined with placebo Respimat® inhaler) twice daily (bid) in the morning and evening for a treatment period of 8 weeks.
Period: Overall Study
Arm/Group | BI 54903 90.9μg Bid | BI 54903 181.8μg Bid | BI 54903 363.6μg Bid | Fluticasone Propionate 88μg Bid | Fluticasone Propionate 440μg Bid
Started | 2 | 2 | 1 | 2 | 2
Completed | 0 | 1 | 0 | 0 | 0
Not Completed | 2 | 1 | 1 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0
Not completed — Withdraw due to trial termination | 2 | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Treated set: The treated set consist of all randomized patients where at least one dose of study medication was taken.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 54903 90.9μg Bid | BI 54903 181.8μg Bid | BI 54903 363.6μg Bid | Fluticasone Propionate 88μg Bid | Fluticasone Propionate 440μg Bid | Total
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.0 (2.8) | 42.5 (12.0) | 48.0 (0) | 51.0 (1.4) | 50.5 (14.8) | 45.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1 | 2 | 4
  Male | 2 | 1 | 1 | 1 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 2 | 1 | 1 | 2 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 0 | 2
  White | 1 | 1 | 1 | 1 | 2 | 6
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Randomisation Baseline to the End of the 8-week Treatment Period in Trough (Morning Pre-dose and Pre-rescue Bronchodilator) Forced Expiratory Volume in One Second (FEV1)
Description: Mean change from randomisation baseline to the end of the 8-week treatment period in trough (morning pre-dose and pre-rescue bronchodilator) Forced expiratory volume in one second (FEV1).
Time Frame: At baseline and week 8
Population: Study was terminated by the decision of sponsor. No valid data for primary and secondary endpoints were collected and no analyses of primary and secondary endpoints were conducted.
Arm/Group | BI 54903 90.9μg Bid | BI 54903 181.8μg Bid | BI 54903 363.6μg Bid | Fluticasone Propionate 88μg Bid | Fluticasone Propionate 440μg Bid
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Mean Changes From Randomization Baseline in Trough (Morning Pre-dose and Pre-rescue Bronchodilator) Forced Vital Capacity (FVC) After 2, 4 and 8-week Treatment Periods
Description: Mean changes from randomization baseline in trough (morning pre-dose and pre-rescue bronchodilator) forced vital capacity (FVC) after 2, 4 and 8-week treatment periods.
Time Frame: At baseline and week 2, 4, 8.
Population: as for outcome 1
Arm/Group | BI 54903 90.9μg Bid | BI 54903 181.8μg Bid | BI 54903 363.6μg Bid | Fluticasone Propionate 88μg Bid | Fluticasone Propionate 440μg Bid
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Mean Changes From Randomization Baseline in Trough (Morning Pre-dose and Pre-rescue Bronchodilator) FEV1 After 2 and 4-week Treatment Periods
Description: Mean changes from randomization baseline in trough (morning pre-dose and pre-rescue bronchodilator) FEV1 after 2 and 4-week treatment periods.
Time Frame: At baseline and week 2 and 4.
Population: as for outcome 1
Arm/Group | BI 54903 90.9μg Bid | BI 54903 181.8μg Bid | BI 54903 363.6μg Bid | Fluticasone Propionate 88μg Bid | Fluticasone Propionate 440μg Bid
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Mean Pre-dose (and Pre-rescue) Peak Expiratory Flow (PEF) as Assessed Via Asthma Monitor2+ (AM2+) in the Morning and Evening of the Last Week of the 8-week Treatment Period
Description: Mean pre-dose (and pre-rescue) peak expiratory flow (PEF) as assessed via Asthma Monitor2+ (AM2+) in the morning and evening of the last week of the 8-week treatment period.
Time Frame: At week 8.
Population: as for outcome 1
Arm/Group | BI 54903 90.9μg Bid | BI 54903 181.8μg Bid | BI 54903 363.6μg Bid | Fluticasone Propionate 88μg Bid | Fluticasone Propionate 440μg Bid
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Mean Rescue Medication Use (Daytime and Night-time) as Assessed Via AM2+ in the Morning and Evening of the Last Week of the 8-week Treatment Period
Description: Mean rescue medication use (daytime and night-time) as assessed via AM2+ in the morning and evening of the last week of the 8-week treatment period.
Time Frame: At week 8.
Population: as for outcome 1
Arm/Group | BI 54903 90.9μg Bid | BI 54903 181.8μg Bid | BI 54903 363.6μg Bid | Fluticasone Propionate 88μg Bid | Fluticasone Propionate 440μg Bid
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Mean Change From Randomisation Baseline in ACQ-6 Scores at Subsequent Study Visits
Description: The Asthma Control Questionnaire (ACQ) consists of 6 patient self-evaluated questions with each question in 7-point scale. The items are equally weighted and the ACQ score is the mean of 6 items and ranges between 0 (well controlled) and 6 (extremely poorly controlled). Mean scores of less than or equal to 0.75 indicate well-controlled asthma, scores between 0.76 and less than 1.5 indicate partly controlled asthma, and a score greater than or equal to 1.5 indicates uncontrolled asthma.
Time Frame: At baseline and week 2, 4, 8.
Population: as for outcome 1
Arm/Group | BI 54903 90.9μg Bid | BI 54903 181.8μg Bid | BI 54903 363.6μg Bid | Fluticasone Propionate 88μg Bid | Fluticasone Propionate 440μg Bid
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Mean Change From Randomisation Baseline in Asthma Quality of Life Questionnaire (AQLQ(S)+12) Scores at Subsequent Study Visits
Description: AQLQ(S)+12 are well established and validated questionnaires to measure control of asthma symptoms and quality of life, which is a patient-reported self-administered outcome questionnaire containing 32 items. Each item is scored on a 7-point scale (1=maximal impairment, 7=no impairment). The 32 items of the questionnaire are averaged to produce one overall quality of life score ranging from 1 (severely impaired) to 7 (not impaired at all). Higher scores indicate better quality of life.
Time Frame: At baseline and week 2, 4, 8.
Population: as for outcome 1
Arm/Group | BI 54903 90.9μg Bid | BI 54903 181.8μg Bid | BI 54903 363.6μg Bid | Fluticasone Propionate 88μg Bid | Fluticasone Propionate 440μg Bid
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Time to Withdrawal Due to First Asthma Exacerbation
Description: Time to withdrawal due to first asthma exacerbation.
Time Frame: At week 8.
Population: as for outcome 1
Arm/Group | BI 54903 90.9μg Bid | BI 54903 181.8μg Bid | BI 54903 363.6μg Bid | Fluticasone Propionate 88μg Bid | Fluticasone Propionate 440μg Bid
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Mean Change From Randomization Baseline in Through (Morning Pre-dose and Pre-rescue Bronchodilator) FEF 25-75 After 2, 4 and 8-week Treatment Periods
Description: Mean change from randomization baseline in through (morning pre-dose and pre-rescue bronchodilator) Forced expiratory flow between 25% and 75% of vital capacity (FEF 25-75) after 2, 4 and 8-week treatment periods.
Time Frame: At baseline and week 2, 4 and 8.
Population: as for outcome 1
Arm/Group | BI 54903 90.9μg Bid | BI 54903 181.8μg Bid | BI 54903 363.6μg Bid | Fluticasone Propionate 88μg Bid | Fluticasone Propionate 440μg Bid
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization until 8 weeks at end of trial + 2 weeks of follow-up period, up to 10 weeks
Description: The treated sets consist of all randomized patients where at least one dose of study medication was taken.
Arm/Group | BI 54903 90.9μg Bid | BI 54903 181.8μg Bid | BI 54903 363.6μg Bid | Fluticasone Propionate 88μg Bid | Fluticasone Propionate 440μg Bid
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/1 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/1 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 0/2 | 0/1 | 2/2 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 54903 90.9μg Bid (N=2) | BI 54903 181.8μg Bid (N=2) | BI 54903 363.6μg Bid (N=1) | Fluticasone Propionate 88μg Bid (N=2) | Fluticasone Propionate 440μg Bid (N=2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Study was terminated by the decision of sponsor. As limited data were collected due to early termination and only limited number of patients completing the 8-week treatment period, no analyses of primary and secondary endpoints were conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.